CLINICAL TRIAL: NCT00002258
Title: A Phase I, Open Label Trial to Evaluate the Safety, Tolerance and Biological Effects of SDZ ILE-964 (Recombinant Human Interleukin-3, RhIL-3) in HIV Infected Patients With Cytopenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 080A; B104
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-11

CONDITIONS: HIV Infections; Cytopenias
Keywords: Interleukin-3; Recombinant Proteins; Leukopenia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Thrombocytopenia
MeSH Terms: conditions — HIV Infections; Cytopenia; Leukopenia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Thrombocytopenia | interventions — Interleukin-3

INTERVENTIONS:
Drug: Interleukin-3

SUMMARY:
To determine the safety, tolerability and maximum tolerated dose of SDZ ILE 964 administered by daily subcutaneous injections in patients infected with human immunodeficiency virus (HIV) who have cytopenias (low blood cell counts). To obtain information about the biologic effects of SDZ ILE 964 administration in improving blood counts in HIV-infected patients. To obtain information about the effects of SDZ ILE-964 administration on both parameters of HIV replication and on residual immunologic function.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity by Western blot.
* Advanced ARC or AIDS as defined by CDC.
* Cytopenia defined as total peripheral leukocyte count of < 3,000 cells/mm3 or platelet count of < 100,000 cells/mm3 or serum hemoglobin < 10 g/dl.
* Anticipated life expectancy = or > 6 months.
* Ambulatory.
* Willing to sign informed consent.
* Willing to forego use of any other investigational therapies except ddI.

Prior Medication:

Allowed > 2 weeks prior to study entry:

* zidovudine.
* Allowed > 4 weeks prior to study entry:
* systemic cytotoxic chemotherapy; investigational drugs; medications known to be myelosuppressive as ganciclovir, trimethoprim/sulfamethoxazole or dapsone.
* Allowed > 6 weeks prior to study entry:
* other hemopoietic growth factor treatment as GM-CSF, EPO.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection.
* Symptoms of CNS disease referable to HIV infection.
* Dementia or altered mental status that would prohibit giving and understanding informed consent.

Systemic chemotherapy.

* Investigational therapies other than ddI.
* Medications with known myelosuppressive effects such as ganciclovir, trimethoprim/sulfamethoxazole or dapsone or AZT.
* Other hematopoietic growth factor treatments as GM-CSF, G-CSF, or EPO.

Prophylactic therapy for pneumocystis or oral thrush.

* ddI.
* Corticosteroids or topical corticosteroid creams.

Patients may not have:

* Life expectancy < 6 months.
* Active drug or alcohol abuse.
* Active opportunistic infections.
* Treatment with any other investigational drugs except ddI within 4 weeks of study entry.
* Dementia or altered mental state that prohibits giving informed consent.
* Symptoms of CNS disease referable to HIV infection.
* Major surgery within 4 weeks of study entry.
* History of major pulmonary or cardiac disease.
* History of any prior malignancy other than Kaposi's sarcoma or noninvasive subcutaneous carcinoma.
* Documented allergic disorder such as asthma, history of anaphylaxis, atopy, serum sickness, or bronchospasm.

Not allowed within 2 weeks prior to study entry:

* zidovudine (AZT).
* Not allowed within 4 weeks prior to study entry:
* systemic cytotoxic chemotherapy; investigational drugs other than ddI; medications known to be myelosuppressive as ganciclovir, trimethoprim/sulfamethoxazole or dapsone.
* Not allowed within 6 weeks prior to study entry:
* other hematopoietic growth factor treatment as GM-CSC, G-CSF, EPO.

Radiation therapy or major surgery within 4 weeks of study entry.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- New England Deaconess Hosp, Boston, Massachusetts, United States

REFERENCES:
- [Background] Scadden DT, Levine JD, Bresnahan J, Gere J, McGrath J, Wang Z, Resta DJ, Young D, Hammer SM. In vivo effects of interleukin 3 in HIV type 1-infected patients with cytopenia. AIDS Res Hum Retroviruses. 1995 Jun;11(6):731-40. doi: 10.1089/aid.1995.11.731. PMID 7576933
- [Background] Levine AM, Li P, Cheung T, Tulpule A, Von Roenn J, Nathwani BN, Ratner L. Chemotherapy consisting of doxorubicin, bleomycin, vinblastine, and dacarbazine with granulocyte-colony-stimulating factor in HIV-infected patients with newly diagnosed Hodgkin's disease: a prospective, multi-institutional AIDS clinical trials group study (ACTG 149). J Acquir Immune Defic Syndr. 2000 Aug 15;24(5):444-50. doi: 10.1097/00126334-200008150-00009. PMID 11035615